CLINICAL TRIAL: NCT06837168
Title: Clinical Effectiveness of Cobalt Chromium CAD-CAM Designed Customized Lingual Retainer: a Randomized Clinical Trial
Brief Title: Clinical Effectiveness of Cobalt Chromium CAD-CAM Designed Customized Lingual Retainer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hiba Muhammed, Principal investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1021425
Record Dates: First submitted 2025-02-03; First posted 2025-02-20 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Tooth Stability; Periodontal Health; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAD/CAM 3D Printed Chrome Cobalt Fixed Retainers group (Active Comparator): The participant will receive a fixed retainer fabricated using computer-aided design and computer-aided manufacturing (CAD/CAM) technology. The retainer will be constructed from cobalt-chromium. The CAD/CAM process involved scanning the patient's dental arch to create a digital model, which was then used to design the retainer. The retainer will be bonded to the lingual surfaces of the mandibular incisors and canines, extending from canine to canine. Participants were instructed to maintain proper oral hygiene and attend regular follow-up appointments.
  Interventions: Device: 3D printed CAD/CAM Chrome cobalt fixed lingual retainers
- Stainless steel Fixed Retainer group (Active Comparator): participants will receive a fixed orthodontic retainer fabricated from a 0.0215-inch, five-stranded stainless steel wire. The retainer will be bonded to the lingual surfaces of the mandibular incisors and canines, extending from canine to canine. Participants were instructed to maintain proper oral hygiene and attend regular follow-up appointments.
  Interventions: Device: Stainless steel fixed retainer

INTERVENTIONS:
Device: Stainless steel fixed retainer — The Stainless steel fixed orthodontic retainer is fabricated from a 0.0215-inch, five-stranded stainless steel wire
  Arms: Stainless steel Fixed Retainer group
Device: 3D printed CAD/CAM Chrome cobalt fixed lingual retainers — CAD/CAM Chrome cobalt retainers; will be digitally designed by the dental technician using EXOCAD software. Then, they will be printed by DMP Flex100 metal 3D printer and then will be polished. Also, a projection like extensions will be added at the ends of the retainers to avoid slippage in addition to gingivally directed V notch shaped bend in the retainer to increase the retention in the anterior region
  Arms: CAD/CAM 3D Printed Chrome Cobalt Fixed Retainers group

SUMMARY:
This study aims to evaluate the clinical effectiveness of CAD/CAM 3D printed Chrome Cobalt fixed retainer in maintaining mandibular anterior teeth stability.

The Research Question; "Does the Cobalt-Chromium CAD/CAM designed customized lingual retainer better than Stainless steel lingual retainer in improving tooth stability after orthodontic treatment?" The null hypothesis "There is no differences between the fixed CAD/CAM 3D printed Chrome Cobalt customized retainer and the multi-stranded stainless-steel fixed retainer in maintaining mandibular anterior teeth stability."

DETAILED DESCRIPTION:
A multicenter, single-blinded, randomized controlled trial will be consist of three main parts:

1. Questionnaire Survey - A cross-sectional survey will be distributed to orthodontists to assess their experience and perception of CAD/CAM retainers.
2. In Vitro Study - Laboratory tests will be performed on different diameters of CAD/CAM cobalt-chromium retainers to evaluate their mechanical properties, including tensile strength, load deflection, and shear bond strength.
3. Clinical trial to to evaluate the effectiveness of CAD/CAM retainer group in minimizing the 6month post-orthodontic treatment change in term of a Little's Irregularity Index (LII).

42 Patients will be enrolled; at the last appointment of orthodontic treatment before debonding, subjects will be assessed for the presence of good gingival health parameters using the BPE. Then the patients will have supra gingival debridement followed by an intraoral scan for lower arch; Intraoral scans will be taken for all the participants and STL files will be generated. In addition, a stone model will be made for the lower arch of the control group.

Group 1 (CAD/CAM retainers): STL files will be sent to lab. Group 2 (conventional retainers): The retainer wire will be shaped to adapt passively to the lingual surfaces of lower anterior teeth on the stone model. A silicone transfer key will be prepared to facilitate the positioning of the retainers Laboratory work: CAD/CAM Chrome cobalt retainers; will be digitally designed by the dental technician using EXOCAD software. Then, they will be 3D printed by metal 3D printer and then will be polished. Also, a projection like extensions will be added at the ends of the retainers to avoid slippage in addition to gingivally directed V notch shaped bend in the retainer to increase the retention in the anterior region.

Bonding procedures: The operators will first check the fitting and adaptation of the retainers on the teeth. After cleaning the teeth and isolate them by placement the rubber dam; 35% phosphoric acid etchant gel will be applied. Bonding agent, as the manufacturer's recommendations will be used, After completing the bonding procedure, the patient will be recalled after one week to measure the parameters of gingival health to exclude the plaque retentive fixed appliance effect. The patient will be given oral hygiene instructions and encouraged to use the interdental brush and will be advised to contact the clinician as soon as possible if they have any concerns or problems.

ELIGIBILITY:
Inclusion Criteria:

* Completion of a course of fixed appliance therapy.
* with a satisfactory correction of malocclusion and dental alignment.
* Class I canine relationship based on Andrew's criteria for finishing.
* Patients with a history of constant oral hygiene measures daily.
* Good general health.
* Subjects had a full and normal complement of teeth in the lower labial segments.
* Teeth within the labial segments should be regularly sized and shaped.
* Subjects willing to consent to the trial.

Exclusion Criteria:

* Patients with a deep overbite
* Patients with traumatic parafunctional habits such as bruxism and clenching.
* Patients with carious, restored, fractured, or missing lower anterior teeth.
* Patients with medical health problems that may influence gingival health, like uncontrolled type II diabetic patients.
* patients under systemic drug administration that affects oral health.
* Smokers

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of CAD/CAM 3D printed Chrome Cobalt fixed retainers | from 1st day of retainer insertion to the last of initial (first ) 6 months of retention
  Evaluate the effectiveness of CAD/CAM 3D printed Chrome Cobalt fixed retainers a in term of post-treatment stability of mandibular anterior teeth over a 6-month period by using Little's Irregularity Index. Post-treatment changes in millimeters will be defined as change in labial segment alignment.

SECONDARY OUTCOMES:
Retainer survival | from 1st day of retainer insertion to the last of initial (first ) 6 months of retention
Patient satisfaction | after 3 months of retainer insertion to the last of initial (first ) 6 months of retention
  the patient experience with the new retainer will be evaluated through the Visual Analogue Scale regarding comfort/satisfaction with the Fixed retainers.
  There will be five questions relating to how comfortable he/she finds the retainers and how they affect the daily life. Each question must be answered by number from 0 to 100; The left side represents 0 = complete satisfaction/comfort The right side represents 100 = complete discomfort/unsatisfaction
inter-canine width | from 1st day of retainer insertion to the last of initial (first ) 6 months of retention
  the distance between cusp tips of right and left mandibular canines in millimeters.
The pattern of wire failure | from 1st day of retainer insertion to the last of initial (first ) 6 months of retention
  The pattern of failure will be recorded:
  the wire-composite interface; the enamel-composite interface; wire fracture; or complete detachment from all teeth
overjet | from 1st day of retainer insertion to the last of initial (first ) 6 months of retention
  The horizontal distance ( in millimeters) between Maxillary incisor edge labial surface of Mandibular incisors
Overbite | from 1st day of retainer insertion to the last of initial (first ) 6 months of retention
  The distance of maximum vertical overlap ( in millimeters) between Maxillary and Mandibular incisors in maximum intercuspation.
assessment of plaque accumulation | after 3 months of retainer insertion to the last of initial (first ) 6 months of retention
  by using plaque- disclosing agent and painting all the surfaces of the teeth Plaque index then calculated.
Periodontal Probing Depth. | after 3 months of retainer insertion to the last of initial (first ) 6 months of retention
  measured in mm using periodontal prob.
Bleeding on Probing | after 3 months of retainer insertion to the last of initial (first ) 6 months of retention

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Ali Mohammed Hameed, Study Director — University of Baghdad
Locations (1):
- University of Baghdad - College of Dentistry, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumrular B, Cicek O, Dag IE, Avar B, Erener H. Evaluation of the Corrosion Resistance of Different Types of Orthodontic Fixed Retention Appliances: A Preliminary Laboratory Study. J Funct Biomater. 2023 Jan 31;14(2):81. doi: 10.3390/jfb14020081. PMID 36826880
- [Background] Cokakoglu S, Adanur-Atmaca R, Cakir M, Ozturk F. Stability and failure rate during 3 years of fixed retention: A follow-up of an randomized clinical trial on adolescents with four different lingual retainers. Orthod Craniofac Res. 2024 Apr;27(2):251-258. doi: 10.1111/ocr.12714. Epub 2023 Oct 3. PMID 37786933
- [Background] Shim H, Foley P, Bankhead B, Kim KB. Comparative assessment of relapse and failure between CAD/CAM stainless steel and standard stainless steel fixed retainers in orthodontic retention patients. Angle Orthod. 2022 Jan 1;92(1):87-94. doi: 10.2319/121720-1015.1. PMID 34464438
- [Background] Gera A, Pullisaar H, Cattaneo PM, Gera S, Vandevska-Radunovic V, Cornelis MA. Stability, survival, and patient satisfaction with CAD/CAM versus conventional multistranded fixed retainers in orthodontic patients: a 6-month follow-up of a two-centre randomized controlled clinical trial. Eur J Orthod. 2023 Feb 10;45(1):58-67. doi: 10.1093/ejo/cjac042. PMID 35964235
- [Background] Alnuaimy NS, Alhuwaizi AF. A Novel 3-Dimensional Printed Nanoceramic Hybrid Resin Fixed Lingual Retainer: Characterization and Mechanical Tests. Int J Dent. 2024 Oct 15;2024:3540846. doi: 10.1155/2024/3540846. eCollection 2024. PMID 39445113
- [Background] ISO.15841, Dentistry-Wires for Use in Orthodontics (Geneva, Switzerland: International Organization for Standardization, 2nd edition, 2014): 5-7.
- [Background] Baysal A, Uysal T, Gul N, Alan MB, Ramoglu SI. Comparison of three different orthodontic wires for bonded lingual retainer fabrication. Korean J Orthod. 2012 Feb;42(1):39-46. doi: 10.4041/kjod.2012.42.1.39. Epub 2012 Feb 27. PMID 23112930